CLINICAL TRIAL: NCT05056727
Title: A Phase 3, International, Randomised, Double-blind, Placebo-controlled Study to Evaluate the Effect of Sodium Zirconium Cyclosilicate on CKD Progression in Participants With CKD and Hyperkalaemia or at Risk of Hyperkalaemia
Brief Title: A Study to Evaluate the Effect of Sodium Zirconium Cyclosilicate on Chronic Kidney Disease (CKD) Progression in Participants With CKD and Hyperkalaemia or at Risk of Hyperkalaemia
Acronym: STABILIZE-CKD
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study started enrollment in Sep 2021 and despite huge efforts the rate of patient enrollment continued to be below target such that the completion of the study within a reasonable timeframe was deemed very unlikely.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9488C00001; 2021-001911-96 (EudraCT Number)
Record Dates: First submitted 2021-09-01; First posted 2021-09-24 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Renal Insufficiency, Chronic; Hyperkalemia
Keywords: Renal Insufficiency, Chronic; Chronic Kidney Diseases; Hyperkalemia
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperkalemia | interventions — sodium zirconium cyclosilicate; Lisinopril; Valsartan; Irbesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sodium Zirconium Cyclosilicate (SZC) (Experimental): SZC 5 g every other day to 15 g once daily + Lisinopril/Valsartan
  Interventions: Drug: Sodium Zirconium Cyclosilicate (SZC); Drug: Lisinopril; Drug: Valsartan; Drug: Irbesartan
- Placebo (Placebo Comparator): Placebo + Lisinopril/Valsartan
  Interventions: Drug: Placebo; Drug: Lisinopril; Drug: Valsartan; Drug: Irbesartan

INTERVENTIONS:
Drug: Sodium Zirconium Cyclosilicate (SZC) — Powder for oral suspension in a sachet. Unit dose strength: 5 or 10 g SZC. Single dose will consist of 1-3 sachets.
  During Initiation Phase:
  * S-K > 5 to ≤ 6.5 mmol/L (measured by L-Lab): Single dose contains 10 g SZC that should be suspended in 45 mL of water. The 10 g SZC single dose should be administered three times daily for up to 72 hours until normokalaemic (S-K 3.5-5.0 mmol/L); the total daily dose is 30 g SZC.
  * S-K ≥ 3.5 to ≤ 5 mmol/L (measured by L-Lab): Single dose contains 5 g SZC that should be suspended in 45 mL of water and administered once daily for 48 hours.
  During Run-in and Maintenance Phases:
  - Single dose contains 5 g SZC administered every other day or 5, 10, or 15 g SZC administered once daily that should be suspended in 45 mL of water.
  Other Names: Lokelma TM
  Arms: Sodium Zirconium Cyclosilicate (SZC)
Drug: Placebo — Powder for oral suspension in a sachet. Placebo to match 5 or 10 g. Single dose will consist of 1-3 sachets.
  During Maintenance Phase:
  - Single dose contains 5 g placebo administered every other day or 5, 10, or 15 g placebo administered once daily that should be suspended in 45 mL of water.
  Arms: Placebo
Drug: Lisinopril — Tablet for oral administration. Unit dose strength: 2.5, 5, 10 or 20 mg. Dosage level: 5, 10, 20, or 40 mg administered once daily.
Drug: Valsartan — Tablet or capsule for oral administration. Unit dose strength: 40, 80 or 160 mg. Dosage level: 40, 80, 160, or 320 mg administered once daily.
Drug: Irbesartan — Tablet for oral administration. Unit dose strength: 75, 150 or 300 mg. Dosage level: 75, 150, or 300 mg administered once daily.
  The study is designed to use valsartan as the selected ARB therapy adjunct to SZC. However, if an actual shortage of valsartan in a local market jeopardises the ability of participants to enter or continue in the study, valsartan can be temporarily substituted with irbesartan until the shortage of valsartan is resolved.

SUMMARY:
The purpose of this study is to evaluate the effect of Sodium Zirconium Cyclosilicate (SZC), as adjunct to ACEi/ARB therapy (lisinopril or valsartan), on slowing CKD progression (assessed as the reduction in participant's glomerular filtration rate [eGFR] decline over time) in participants with hyperkalaemia or at high risk of hyperkalaemia.

DETAILED DESCRIPTION:
This is a Phase 3, international, randomised withdrawal, double-blind, parallel-group, placebo-controlled study, to evaluate the effect of SZC as adjunct to RAASi therapy (lisinopril or valsartan) in slowing CKD progression in participants with CKD and hyperkalaemia or at risk of hyperkalaemia.

Specifically, the study will include participants with hyperkalaemia (S-K > 5.0 to ≤ 6.5 mmol/L by central laboratory) who are on adequate or limited RAASi therapy due to hyperkalaemia, and participants with normokalaemia (S-K ≥ 3.5 to ≤ 5.0 mmol/L by central laboratory) who are on limited RAASi therapy due to high risk of hyperkalaemia. High risk of hyperkalaemia is defined as (1) participants with a previous medical history or record of hyperkalaemia within the prior 24 months who are on limited RAASi therapy despite indication in CKD; (2) participants in whom RAASi therapy is indicated in CKD but are on limited RAASi therapy and have S-K ≥ 4.7 to ≤ 5.0 mmol/L; and (3) participants in whom RAASi therapy has been discontinued or reduced to suboptimal doses because of hyperkalaemia.

A participant is expected to be in the study for approximately 28 months, which includes up to 13 days for the screening period, 27 months for the intervention period, and 1 week for follow-up. The 27-month intervention period of the study consists of 3 phases, an initiation phase (up to 72 hours), a run-in phase (3 months/up to Day 90), and a maintenance phase (24 months/104 weeks).

The initial dose of SZC will be administered to participants during the initiation phase. No changes will be made to the ACEi or ARB therapy at this stage. As soon as possible after the participant is confirmed to be normokalaemic at the end of the initiation phase, the participant will enter the run-in phase. Participants will receive open-label SZC and either lisinopril or valsartan. The aim of the run-in phase is to increase ACEi or ARB therapy stepwise to their maximum doses. After a 3-month run-in period for RAASi dose optimization while on SZC, participants will be randomized to SZC or placebo and followed during the subsequent 24 months of maintenance phase for efficacy and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and protocol
* Must be ≥ 18 years of age at the time of signing the informed consent.
* Must have eGFR ≥ 25 and ≤ 59 mL/min/1.73m2 as calculated by central laboratory (CKD-EPI formula) at screening (Visit 1)
* Must have UACR ≥ 200 and ≤ 5000 mg/g as calculated by central laboratory at screening (Visit 1). If the first sample does not fulfil eligibility criteria, a second sample can be obtained during the screening period; if so, the UACR measurement from the second sample must be within the eligibility range.
* Any of the following criteria, a or b, at screening (Visit 1):

  1. Cohort A: Hyperkalaemia (S-K > 5.0 to ≤ 6.5 mmol/L) as measured by the central laboratory, and on adequate* or limited** RAASi therapy due to hyperkalaemia.
  2. Cohort B: Normokalaemia (S-K ≥ 3.5 to ≤ 5.0 mmol/L) as measured by the central laboratory and on limited** RAASi therapy due to high risk of hyperkalaemia. High risk of hyperkalaemia is defined as:

  (i) Participants with a previous medical history or record of hyperkalaemia within the prior 24 months, who are on limited** RAASi therapy despite indication in CKD.

(ii) Participants in whom RAASi therapy is indicated in CKD, who are on limited** RAASi therapy and have S-K ≥ 4.7 to ≤ 5.0 mmol/L.

(iii) Participants in whom RAASi therapy has been discontinued or reduced to suboptimal* doses because of hyperkalaemia.

*Adequate RAASi dose levels are defined in protocol; doses lower than these are considered as suboptimal.

**Limited RAASi therapy is defined as no or suboptimal RAASi therapy according to dosing guidance provided in protocol.

* If on thiazide or loop diuretics, the dose must have been stable for 2 weeks prior to screening (Visit 1).
* If on RAASi therapy, the dose must have been stable for one month prior to screening (Visit 1) and remain stable during screening.
* If on an SGLT2i treatment (ie, dapagliflozin and canagliflozin), finerenone, or any other medications in these 2 classes that are approved for CKD, the dose must have been stable for 3 months prior to screening (Visit 1).
* Participants must be one-year postmenopausal, surgically sterile, or using one highly effective form of birth control (defined as one that can achieve a failure rate of less than 1% per year when used consistently and correctly). They should have been stable on their chosen method of birth control for a minimum of one month prior to screening (Visit 1) and willing to remain on the birth control until one month after the last dose of study intervention.

Exclusion Criteria:

* New York Heart Association class III to IV congestive heart failure at the time of screening (Visit 1) or previous history of severe or symptomatic heart failure.
* Myocardial infarction, unstable angina, stroke, or transient ischaemic attack within 3 months prior to screening (Visit 1).
* Participants with a known history of systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 95 mmHg within 2 weeks prior to screening (Visit 1) are excluded. In addition, any participant with systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 95 mmHg as measured at screening (Visit 1) and confirmed by repeated measurement is excluded. Participants may be rescreened once blood pressure is controlled.
* QTcF > 550 msec at screening (Visit 1).
* History of QT prolongation associated with other medications that required discontinuation of that medication.
* Congenital long QT syndrome.
* Symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia. Participants with atrial fibrillation and heart rate controlled by medication are permitted.
* Lupus nephritis or anti-neutrophil cytoplasmic antibody-associated vasculitis.
* Change in renal function requiring hospitalisation or dialysis within 3 months prior to screening (Visit 1).
* History of renal transplant (or anticipated need for renal transplant during the study).
* Severe hepatic impairment, biliary cirrhosis, or cholestasis.
* History of hereditary or idiopathic angioedema.
* Any prior hypersensitivity to ACEi or ARB that in the investigator's judgment precludes use of lisinopril and valsartan/irbesartan. Prior hypersensitivity reactions to consider include, but are not limited to, development of angioedema, icterus, hepatitis, or neutropaenia or thrombocytopaenia requiring treatment modification.
* Known hypersensitivity or previous anaphylaxis to SZC or to components thereof.
* Any condition outside the CV and renal disease area such as, but not limited to, malignancy, with a life expectancy of less than 2 years based on investigator´s clinical judgment.
* Active malignancy requiring treatment at the time of screening (Visit 1), except for successfully treated basal cell or treated squamous cell carcinoma.
* S-K > 6.5 or < 3.5 mmol/L by local laboratory within 1 day prior to the scheduled first dose of SZC in the initiation phase.
* Evidence of COVID-19 infection within 2 weeks prior to screening (Visit 1).
* Treated with dual blockade of RAAS (combined use of an ACEi and ARB) within 3 months prior to screening (Visit 1).
* Treated with an angiotensin receptor neprilysin inhibitor (ARNI; sacubitril/valsartan [Entresto®]) within 3 months prior to screening (Visit 1).
* Treated with an MRA not approved for CKD within 3 months prior to screening (Visit 1).
* Treated with aliskiren-containing products with 3 months prior to screening (Visit 1).
* Treated with SPS (eg, Kayexalate, Resonium), CPS (Resonium Calcium), patiromer (Veltassa®), or SZC (Lokelma®) within 7 days prior to screening (Visit 1).
* Participation in another clinical study with an investigational product administered within one month prior to screening (Visit 1).
* Not willing or not able to change to lisinopril or valsartan/irbesartan, the protocol-mandated RAASi study intervention. Note: For participants taking a fixed combination of an ACEi or ARB with another agent (eg, calcium blockers or diuretics) as SoC, the investigator must make a judgment that it will be safe and efficacious for such participants to change to the study ACEi or ARB and to the other drug as separate agents.
* Previous dosing with SZC in the present study.
* Currently pregnant (confirmed with positive pregnancy test at screening [Visit 1]) or breastfeeding.
* Judgment by the investigator that the participant is unlikely to comply with study procedures, restrictions, and requirements.
* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1112 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2024-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn M. Chertow, MD, MPH, Principal Investigator — Stanford University School of Medicine, Stanford, CA USA
Locations (223):
- United States (39):
  - Research Site, Surprise, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Canyon Country, California
  - Research Site, Chula Vista, California
  - Research Site, Northridge, California
  - Research Site, San Dimas, California
  - Research Site, South Gate, California
  - Research Site, Tarzana, California
  - Research Site, Denver, Colorado
  - Research Site, Boynton Beach, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Ocoee, Florida
  - Research Site, Temple Terrace, Florida
  - Research Site, Nampa, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Oak Brook, Illinois
  - Research Site, Fort Wayne, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Flint, Michigan
  - Research Site, Saint Clair Shores, Michigan
  - Research Site, Columbia, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Albuquerque, New Mexico
  - Research Site, Albany, New York
  - Research Site, Great Neck, New York
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Chester, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Newport News, Virginia
- Argentina (7):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, Rosario
  - Research Site, San Vicente
  - Research Site, Sarandí
- Brazil (6):
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Joinville
  - Research Site, Maringá
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Bulgaria (16):
  - Research Site, Blagoevgrad
  - Research Site, Botevgrad
  - Research Site, Dupnitsa
  - Research Site, Gorna Oryahovitsa
  - Research Site, Gotse Delchev
  - Research Site, Kozloduy
  - Research Site, Lom
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Samokov
  - Research Site, Sandanski
  - Research Site, Silistra
  - Research Site, Sliven
  - Research Site, Smolyan
  - Research Site, Stara Zagora
  - Research Site, Yambol
- Canada (3):
  - Research Site, Saint John, New Brunswick
  - Research Site, Oshawa, Ontario
  - Research Site, Montreal, Quebec
- China (32):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Hengyang
  - Research Site, Huizhou
  - Research Site, Lanzhou
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Sanya
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shengyang
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Taiyuan
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Xuzhou
  - Research Site, Yantai
  - Research Site, Yinchuan
  - Research Site, Zhengzhou
  - Research Site, Zhuzhou
- India (4):
  - Research Site, Coimbatore
  - Research Site, Kolkata
  - Research Site, Madurai
  - Research Site, New Delhi
- Italy (10):
  - Research Site, Bari
  - Research Site, Bassano del Grappa
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Messina
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Rozzano
  - Research Site, San Giovanni Rotondo
  - Research Site, Verona
- Japan (37):
  - Research Site, Amagasaki-shi
  - Research Site, Atsugi-shi
  - Research Site, Chiba
  - Research Site, Chuo-shi
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Kamakura-shi
  - Research Site, Kanoya-shi
  - Research Site, Kasugai-shi
  - Research Site, Kawachinagano-shi
  - Research Site, Kawasaki-shi
  - Research Site, Kitakyushu
  - Research Site, Kitakyushu-shi
  - Research Site, Koriyama-shi
  - Research Site, Koshigaya-shi
  - Research Site, Kumamoto
  - Research Site, Kure-shi
  - Research Site, Marugame-shi
  - Research Site, Matsumoto-shi
  - Research Site, Matsusaka-shi
  - Research Site, Matsuyama
  - Research Site, Nagoya
  - Research Site, Naka
  - Research Site, Noda
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Ōmihachiman
  - Research Site, Sakaishi
  - Research Site, Takarazuka-shi
  - Research Site, Toyota
  - Research Site, Toyota-Shi
  - Research Site, Tsu
  - Research Site, Tsuchiura-shi
  - Research Site, Urayasu-shi
  - Research Site, Yaizu-shi
  - Research Site, Yokohama
  - Research Site, Yonago-shi
- Malaysia (6):
  - Research Site, Alor Star
  - Research Site, Batu Caves
  - Research Site, Johor Bahru
  - Research Site, Kajang
  - Research Site, Kuala Lumpur
  - Research Site, Seri Manjung
- Mexico (8):
  - Research Site, Cuauhtémoc
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, Mazatlán
  - Research Site, Mérida
  - Research Site, México
  - Research Site, San Luis Potosí City
  - Research Site, Veracruz
- Philippines (2):
  - Research Site, Davao City
  - Research Site, Iloilo City
- Poland (5):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Tczew
- Research Site, Ponce, Puerto Rico
- Russia (5):
  - Research Site, Aramil
  - Research Site, Moscow
  - Research Site, Perm
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
- Spain (9):
  - Research Site, Almería
  - Research Site, Barcelona
  - Research Site, Getafe
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Santa Cruz de Tenerife
  - Research Site, Seville
  - Research Site, Valencia
- Taiwan (8):
  - Research Site, Hualien City
  - Research Site, Kaohsiung City
  - Research Site, Keelung
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chaingmai
  - Research Site, Hat Yai
  - Research Site, Ratchathewi
- Turkey (Türkiye) (9):
  - Research Site, Adapazarı
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Gaziantep
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kahramanmaraş
  - Research Site, Kayseri
  - Research Site, Kocaeli
- Ukraine (7):
  - Research Site, Dnipropetrovsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
  - Research Site, Zhytomyr
- Vietnam (5):
  - Research Site, Biên Hòa
  - Research Site, Da Nang
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Huế

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9488C00001&attachmentIdentifier=bd5e1df8-8d76-4c2b-85a1-868ee6fe9577&fileName=D9488C00001_redacted_CSP.pdf&versionIdentifier=
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9488C00001&attachmentIdentifier=51dfd5ca-876f-4a93-9cb3-e4348f288681&fileName=D9488C00001_redacted_SAP.pdf&versionIdentifier=
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D9488C00001&attachmentIdentifier=d9623d06-218e-49e9-bbae-f27bfc682487&fileName=D9488C00001_Redacted_CSR_Synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 30 September 2021 to 07 February 2024 at 286 sites in 20 countries worldwide.
Pre-assignment Details: 1112 participants entered the initiation phase of the study. 1049 of those participants entered the run-in phase of the study, and a total of 716 participants were randomized to treatment or placebo in the maintenance phase.
Groups:
- Initiation Phase: Initiation phase only:
  5 g SZC QD or 10 g SZC TID
- Run-in Phase: Run-in phase only:
  5 g SZC QOD to 15 g SZC QD, + Lisinopril/Valsartan
- Maintenance Phase: SZC: Maintenance phase only:
  5 g SZC QOD to 15 g SZC QD, + Lisinopril/Valsartan
- Maintenance Phase: Placebo: Maintenance phase only:
  Placebo (for SZC), + Lisinopril/Valsartan
Period: Initiation Phase
Arm/Group | Initiation Phase | Run-in Phase | Maintenance Phase: SZC | Maintenance Phase: Placebo
Started | 1112 (2463 subjects were screened, 1351 were not eligible for Initiation phase.) | 0 | 0 | 0
Completed | 1078 | 0 | 0 | 0
Not Completed | 34 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Study-specific; Study terminated; Other | 20 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0 | 0
Period: Run-in Phase
Arm/Group | Initiation Phase | Run-in Phase | Maintenance Phase: SZC | Maintenance Phase: Placebo
Started | 0 | 1049 (1078 participants completed Initiation phase, 29 were not eligible for Run-in phase.) | 0 | 0
Completed | 0 | 763 | 0 | 0
Not Completed | 0 | 286 | 0 | 0
Not completed — Study-specific; Site terminated; Screen failure; Study terminated; Other | 0 | 237 | 0 | 0
Not completed — Death | 0 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 25 | 0 | 0
Not completed — Physician Decision | 0 | 20 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Period: Maintenance Phase
Arm/Group | Initiation Phase | Run-in Phase | Maintenance Phase: SZC | Maintenance Phase: Placebo
Started | 0 | 0 | 361 (763 participants completed Run-in phase, 47 not eligible for Maintenance phase, 361 randomised to SZC, 359 dosed) | 355 (763 participants completed Run-in phase, 47 not eligible for Maintenance phase, 355 randomised to Placebo, 355 dosed)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 361 | 355
Not completed — Site terminated; Study terminated; Other | 0 | 0 | 332 | 314
Not completed — Withdrawal by Subject | 0 | 0 | 19 | 21
Not completed — Physician Decision | 0 | 0 | 4 | 16
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2
Not completed — Death | 0 | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maintenance Phase: SZC | Maintenance Phase: Placebo | Total
Number analyzed (Participants) | 361 | 355 | 716
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (12.3) | 63.6 (11.9) | 64.0 (12.1)
Age, Customized [Number; unit: Participants]
  18 yr ≤ Age < 65 yr | 163 | 168 | 331
  Age ≥ 65 yr | 198 | 187 | 385
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 132 | 254
  Male | 239 | 223 | 462
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 65 | 79 | 144
  Not Hispanic or Latino | 296 | 276 | 572
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 140 | 133 | 273
  Black or African American | 12 | 13 | 25
  White | 193 | 192 | 385
  Other | 12 | 14 | 26
  Unknown or Not Reported | 4 | 3 | 7
UACR [Median (Inter-Quartile Range); unit: mg/g] — Urine albumin-to-creatinine ratio (UACR); mass concentration of albumin divided by mass concentration of creatinine, in urine.
  Last value within 5 days before first day of Maintenance phase. Population: Full analysis set, participants with a non-missing value.
  mg/g
    number analyzed (Participants) | 354 | 347 | 701
    (all) | 1032.5 [419.0 to 2119.0] | 1017.0 [440.0 to 2056.0] | 1018.0 [439.0 to 2088.0]
eGFR [Mean (Standard Deviation); unit: mL/min/(1.73 m2)] — Estimated glomerular filtration rate (eGFR); formula according to Delgado et al 2022 and Inker et al 2021. Last value within 5 days before first day of Maintenance phase. Population: Full analysis set, participants with a non-missing value.
  mL/min/(1.73 m2)
    number analyzed (Participants) | 348 | 347 | 695
    (all) | 41.0 (12.9) | 40.4 (12.4) | 40.7 (12.6)
S-K [Mean (Standard Deviation); unit: mmol/L] — Serum-potassium (S-K), amount-of-substance concentration of potassium in serum. Central laboratory. Last value within 5 days before first day of Maintenance phase. Population: Full analysis set, participants with a non-missing value.
  mmol/L
    number analyzed (Participants) | 348 | 348 | 696
    (all) | 4.41 (0.43) | 4.45 (0.48) | 4.43 (0.46)

OUTCOME MEASURES:

1. Primary Outcome: Total eGFR Slope (Coprimary Analysis #1)
Description: Total eGFR slope, Baseline (Maintenance phase) to visit 17 (week 69)
Time Frame: Baseline (Maintenance phase) to visit 17 (week 69)
Population: Full analysis set.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/(1.73 m2)/yr
Arm/Group | Maintenance Phase: SZC | Maintenance Phase: Placebo
Number analyzed (Participants) | 352 | 346
mL/min/(1.73 m2)/yr | -5.2975 [-6.6854 to -3.9097] | -4.5622 [-5.9969 to -3.1275]
Statistical Analysis 1: Comparison: Maintenance Phase: SZC vs Maintenance Phase: Placebo; Test type: Other; p = 0.4691, Mixed Models Analysis — Test of no treatment difference in mean total eGFR-slope; Treatment difference in mean slope = -0.7354, 95% CI 2-sided [-2.7311 to 1.2604] — SZC minus Placebo

2. Primary Outcome: Chronic eGFR Slope (Coprimary Analysis #2)
Description: Chronic eGFR slope, 12 weeks to visit 17 (week 69)
Time Frame: 12 weeks to visit 17 (week 69)
Population: Full analysis set.
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/min/(1.73 m2)/yr
Arm/Group | Maintenance Phase: SZC | Maintenance Phase: Placebo
Number analyzed (Participants) | 352 | 346
mL/min/(1.73 m2)/yr | -4.8705 [-6.7222 to -3.0189] | -2.8285 [-4.7571 to -0.8999]
Statistical Analysis 1: Comparison: Maintenance Phase: SZC vs Maintenance Phase: Placebo; Test type: Other — Test of no treatment difference in mean chronic eGFR slope; p = 0.1338, Mixed Models Analysis; Treatment difference in mean slope = -2.0421, 95% CI 2-sided [-4.7156 to 0.6314] — SZC minus Placebo

3. Secondary Outcome: Incidence of the Composite of Kidney Failure Outcomes
Description: Incidence of the composite of kidney failure outcomes comprising: sustained ≥ 40% decline in eGFR, onset of ESKD, and death from kidney failure is analyzed based on Cox regression model. Patients with no events are censored at end of maintenance phase or premature discontinuation.
Time Frame: From Baseline (Maintenance phase) up to week 97 (Maintenance phase)
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase: SZC | Maintenance Phase: Placebo
Number analyzed (Participants) | 359 | 354
Participants | 7 | 4
Statistical Analysis 1: Comparison: Maintenance Phase: SZC vs Maintenance Phase: Placebo; Test type: Other — Test of treatment HR = 1; p = 0.390, Regression, Cox; Hazard Ratio (HR) = 1.72, 95% CI 2-sided [0.50 to 5.90] — SZC relative to Placebo

4. Secondary Outcome: Incidence of RAASi Reduction
Description: Incidence of RAASi (lisinopril/valsartan) dose decrease is analyzed based on Cox regression model. Patients with no events are censored at end of maintenance phase or premature discontinuation.
Time Frame: From Baseline (Maintenance phase) up to week 97 (Maintenance phase)
Population: Full analysis set. Subjects on Valsartan/Lisinopril (RAASi) at randomisation.
Measure: Count of Participants; unit: Participants
Arm/Group | Maintenance Phase: SZC | Maintenance Phase: Placebo
Number analyzed (Participants) | 359 | 354
Participants | 55 | 128
Statistical Analysis 1: Comparison: Maintenance Phase: SZC vs Maintenance Phase: Placebo; Test type: Other — Test of treatment HR = 1; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.34, 95% CI 2-sided [0.25 to 0.47] — SZC relative to Placebo

5. Secondary Outcome: UACR
Description: Urine albumin-to-creatinine ratio (UACR); mass concentration of albumin divided by mass concentration of creatinine, in urine; at visit 13 (week 24)
Time Frame: At visit 13 (week 24)
Population: Full analysis set.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/g
Arm/Group | Maintenance Phase: SZC | Maintenance Phase: Placebo
Number analyzed (Participants) | 202 | 190
mg/g | 1513.07 [1253.89 to 1772.24] | 1211.94 [943.14 to 1480.74]
Statistical Analysis 1: Comparison: Maintenance Phase: SZC vs Maintenance Phase: Placebo; Test type: Other — Test of zero treatment difference; p = 0.034, Regression, Linear; Mean Difference = 301.1, 95% CI 2-sided [23.15 to 579.11] — SZC minus Placebo

ADVERSE EVENTS:
Time Frame: Visit 2 - Day 1 (Initiation Phase) up to Visit 20 - Week 97 (Maintenance Phase)
Arm/Group | Initiation Phase | Run-in Phase | Maintenance Phase: SZC | Maintenance Phase: Placebo
All-Cause Mortality (participants affected / at risk) | 0/1112 | 3/1049 | 4/359 | 2/355
Serious Adverse Events (participants affected / at risk) | 0/1112 | 56/1049 | 66/359 | 42/355
Other Adverse Events (participants affected / at risk) | 12/1112 | 221/1049 | 106/359 | 120/355
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initiation Phase (N=1112) | Run-in Phase (N=1049) | Maintenance Phase: SZC (N=359) | Maintenance Phase: Placebo (N=355)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive cerebrovascular disease (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (2) | 5 (5) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vertigo cns origin (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 6 (8) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Glomerulonephritis membranous (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acquired hydrocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (4) | 3 (3) | 1 (3)
Hypertensive urgency (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Granuloma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Emphysematous cholecystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pasteurella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 4 (4) | 4 (4) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (2) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initiation Phase (N=1112) | Run-in Phase (N=1049) | Maintenance Phase: SZC (N=359) | Maintenance Phase: Placebo (N=355)
Hypertension (Vascular disorders) | 0 (0) | 48 (52) | 18 (19) | 13 (15)
Hypotension (Vascular disorders) | 0 (0) | 18 (21) | 12 (12) | 7 (8)
Constipation (Gastrointestinal disorders) | 3 (3) | 30 (30) | 11 (11) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 14 (14) | 12 (12) | 7 (7)
Oedema peripheral (General disorders) | 2 (2) | 38 (41) | 18 (21) | 6 (8)
Covid-19 (Infections and infestations) | 0 (0) | 15 (15) | 12 (12) | 8 (8)
Nasopharyngitis (Infections and infestations) | 1 (1) | 7 (9) | 11 (14) | 6 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 16 (20) | 23 (30) | 93 (119)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 82 (94) | 44 (58) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to recruitment challenges (not safety concerns). The ensuing small number of fully evaluable subjects (716 randomized vs planned 1360) and short follow up (mean 8 - 9 months vs planned 24 months) had a heavy negative impact on the formal statistical analyses, especially slope analyses, and therefore preclude any meaningful conclusions on eGFR slopes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT05056727/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT05056727/SAP_001.pdf